CLINICAL TRIAL: NCT05327478
Title: Direct Comparison of NRP With DHOPE and COR-NMP to Maximize the Use of ECD After DCD Donation in the Netherlands
Brief Title: NRP vs DHOPE vs COR-NMP in ECD-DCD Donation
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jeroen de Jonge, Principal Investigator, head of liver perfusion programme, Erasmus Medical Center
Other Study IDs: EMC-NRP2-2022
Record Dates: First submitted 2022-02-24; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Liver Transplant; Organ Perfusion; Complication of Surgical Procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non ECD: 50-60 years old AND non ECD
  Interventions: Procedure: NRP; Procedure: DHOPE
- ECD: >60 years old or ECD
  Interventions: Procedure: NRP; Procedure: DHOPE; Procedure: COR-NMP

INTERVENTIONS:
Procedure: NRP — Normothermic Regional Perfusion
Procedure: DHOPE — Dual Hypothermic Oxygenated Perfusion
Procedure: COR-NMP — Controlled Oxygenated Rewarming Normothermic Machine Perfusion
  Groups: ECD

SUMMARY:
There is still a discrepancy between the number of liver transplant candidates and the availability of liver grafts, resulting in waiting list mortality. To increase the supply of suitable liver grafts, extended-donor criteria allografts can be used. However, in the case of donation after cardiac death this is not without a risk. Donor after cardiac death (DCD) grafts have increased risk of primary non function and biliary complications, resulting in either retransplantation, patient morbidity or patient death. Due to uncertainty of their quality DCD grafts can be discarded. However, normothermic machine perfusion (NRP) has the potential to overcome these disadvantages of DCD liver grafts. In DCD livers the physiological abdominal circulation is simulated with in vivo, normothermic, oxygenated perfusion during the first two hours after cardiac death. With this perfusion technique, early ischemia can be reversed, surgical damage due to a hasty procedure can be prevented and organs can be tested on viability. In many countries, NRP is obligatory, however this is not the current golden standard in the Netherlands. The primary objective of this study is the utilization of livers after NRP. Secondary study parameters are reasons for graft discard or rejection at proposal, patient- and graft survival, biliary complications, cost assessment of NRP and outcomes of kidney and pancreas transplants. This multicenter, observational study will be performed on adult liver transplant recipients who have been allocated a DCD liver graft (Maastricht type III and V) of a donor above fifty years old. According to current national procurement protocol, grafts procured in region west will be retrieved with NRP followed by dual hypothermic oxygenated perfusion (DHOPE). Grafts retrieved in region East/North will be retrieved using standard rapid retrieval followed by DHOPE, if the donor is aged 50-60. Grafts from donors aged above 60 will undergo controlled oxygenated rewarming normothermic machine perfusion (COR-NMP) after DHOPE.

DETAILED DESCRIPTION:
The persistent discrepancy between the number of patients awaiting liver transplant and the availability of liver grafts. In the Netherlands, still, 1 in 5 either dies on the waiting list or is removed from the waiting list due to deterioration of the disease. To increase the supply of suitable liver grafts, extended-donor criteria allografts can be used. Extended criteria donors (ECD) include older donors, donors with fatty livers, donors with high transaminase levels and donor after circulatory death (DCD). However, because of an inevitable longer period of warm ischemia, DCD livers have increased risk of primary non function and biliary complications, resulting in either patient morbidity, re-transplantation or patient death. Due to uncertainty of the effect of the longer ischemia time on their quality, DCD grafts can be accepted with reluctance or even discarded.

The persistent organ shortage has forced transplant programs to explore options to expand the organ supply. Parallel to this, interest in use of extended criteria donors (ECD) livers drove an evolution in current technique to retrieve, preserve and improve livers before transplantation. Before the era of perfusion, the organs were retrieved by using standard rapid retrieval (SRR) and preserved by static cold storage (SCS). In 1930 researchers have explored machine perfusion as a technique to preserve organs, but nowadays this technique has many more potentials including testing and improving. Currently, there is a wide diversity in different perfusion techniques, varying from in vivo to ex vivo and hypothermic (8-12°C) to normothermic (35-37°C). The rationale behind perfusion is to restore the flow through the organs with a pump to provide oxygen and drugs.

In normothermic regional perfusion (NRP) the physiological abdominal circulation is simulated with in vivo, normothermic, oxygenated perfusion during the first two hours after circulatory death. NRP replaces SRR, because this techniques allows a surgeon to retrieve the organs in a longer timeframe during this perfusion. Also, NRP can reverse early ischemia, reduce ischemic type biliary lesions, prevent surgical damage due to a more relax operation and the potential to test organs. The possibility to test the organ during NRP enables a save environment to transplant livers from older DCD donors above 60 years old. , In many countries, NRP is obligatory in DCD donation, however this is not the current golden standard in the Netherlands. Only in the Dutch Western region the livers of donors after circulatory death (Maastricht type III and V) above 50 years old will undergo NRP.

Independently of age or region, all DCD livers in the Netherlands will undergo dual hypothermic oxygenated perfusion (DHOPE) in the receiving hospital. DHOPE is a dual (through both portal vein and hepatic artery) hypothermic, ex vivo, machine perfusion technique, which depends on the presence of sufficient oxidative mitochondrial metabolism.

subsequentially, oxygenated mitochondria metabolize due to ischemia accumulated succinate and recharge adenosine tri-phosphate, which leads to less reactive oxygen species, less danger signaling and to reduced overall downstream inflammation during later normothermic reperfusion at implantation. , In comparison with SCS, DHOPE has a significant reduction in postreperfusion syndrome, early allograft dysfunction, and non-anastomotic strictures after DCD. For this reason, this perfusion technique is incorporated in the Dutch national protocol for all DCD liver grafts and financed by personal health insurances. High risk donor livers or livers from donors above sixty years old in the Northeastern region will additionally undergo controlled oxygenated rewarming normothermic machine perfusion (COR-NMP) after DHOPE. Normothermic ex vivo machine perfusion has the opportunity to test ECD grafts before transplant. The controlled oxygenated rewarming prevents sudden temperature shifts and subsequentially reduces ischemia reperfusion injury.

The above mentioned techniques with either cold or warm perfusion serve two different goals: cold perfusion (DHOPE) prevents cholangiopathy and warm perfusion (NMP/NRP) can provide a testing area for the organ. Considering two promising warm perfusion techniques, in 2021 the new national protocol was written were NRP was performed in the west and NMP in the northeastern region. To distinguish the differences between these techniques, all the outcomes should be registered. The question remains if NRP and COR-NMP are comparable to each other in patient outcome graft- and patient survival. If these technique are equivalent in outcomes, this techniques can be distinguished based on other characteristics such as utility, cost effectiveness and influence on other organs. The definition of utility is very broad, but in this registration utilization is defined as the offer of a liver from a transplant coordinator to a successful transplant. One other characteristic to distinguish between the different forms of perfusion is cost-effectiveness. NRP may be more cost-effective than NMP since multiple organs are perfused in one procedure, which could potentially also be beneficial for the other perfused organs. As NRP also perfuses other organs, the question remains how this organs respond on this perfusion technique. For kidneys there is evidence that graft survival is similar after donation after brain death (DBD), NRP and SRR.4 The pancreas will not be transplanted after NRP, but in some cases the pancreas can be used for island isolation.

In the context of a wide variety of different perfusion techniques in one small country, the data of these different perfusion techniques are urgently needed to improve procurement, graft outcome and preservation strategies.

ELIGIBILITY:
Inclusion criteria:

* DCD donor (Maastricht type III and V)
* Age above 50 years old and below 75 years old

Exclusion criteria:

* Malignancy (except for primary non-metastatic central nervous system tumors, non-melanoma skin tumors or cured malignancies)
* Active infection (sepsis, meningitis, human immune deficiency virus, rubella, rabies, herpes zoster, tuberculosis)
* Intravenous drug abuse
* Unknown cause of death
* In the case of a NRP procedure: donors with a BMI above 35 and transaminases above 1000 U/I and not decreasing prior to donation are excluded

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potential DCD (Maastricht type III and V) donors above 50 years old and below 75 years old are screened for participation in the national protocol.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Organ utilization rate in percentage | 01-01-2022 to 01-05-2023
  Number of transplanted organs divided by number offered organs
Survival in days | 1 year post transplantation
  Patient and graft survival
Cost effectiveness in difference between treatments in euro's | One year post transplantation
  All medical costs resulting from treatment

SECONDARY OUTCOMES:
Cumulative complications summarized by the comprehensive complication index (CCI) | One year post transplantation
  Complications will be ranked by the CCI
Number of patients with Ischemic cholangiopathy (IC) and anastomotic strictures (AS) | One year post transplantation
  IC is also referred to as non-anastomotic strictures (NAS) or ischemic type biliary lesions (ITBL). IC is defined as a symptomatic patient (e.g., jaundice or cholangitis) with radiological proven irregularity or lumen narrowing in the intra- or extrahepatic donor bile duct in absence of hepatic artery thrombosis. Isolated strictures at the anastomosis are anastomotic strictures.
Length of stay | During peritransplant admission, up to discharge.
  Length of stay in the hospital during the peritransplant admission, measured in days after the transplantation excluding readmission. Also, length of stay on the intensive care unit during the peritransplant admission, including readmission.
Number of patients with Early allograft dysfunction (EAD) | Post operative day 90
  EAD is defined as patient or graft death before the post-operative day (POD) 90
Waiting list time in days | 01-01-2022 to 01-05-2023
  Per center
Waitlist mortality in percentage | 01-01-2022 to 01-05-2023
  Per center

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen de Jonge, Dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Vries Y, Matton APM, Nijsten MWN, Werner MJM, van den Berg AP, de Boer MT, Buis CI, Fujiyoshi M, de Kleine RHJ, van Leeuwen OB, Meyer P, van den Heuvel MC, de Meijer VE, Porte RJ. Pretransplant sequential hypo- and normothermic machine perfusion of suboptimal livers donated after circulatory death using a hemoglobin-based oxygen carrier perfusion solution. Am J Transplant. 2019 Apr;19(4):1202-1211. doi: 10.1111/ajt.15228. Epub 2019 Jan 23. PMID 30588774
- [Background] van Rijn R, Schurink IJ, de Vries Y, van den Berg AP, Cortes Cerisuelo M, Darwish Murad S, Erdmann JI, Gilbo N, de Haas RJ, Heaton N, van Hoek B, Huurman VAL, Jochmans I, van Leeuwen OB, de Meijer VE, Monbaliu D, Polak WG, Slangen JJG, Troisi RI, Vanlander A, de Jonge J, Porte RJ; DHOPE-DCD Trial Investigators. Hypothermic Machine Perfusion in Liver Transplantation - A Randomized Trial. N Engl J Med. 2021 Apr 15;384(15):1391-1401. doi: 10.1056/NEJMoa2031532. Epub 2021 Feb 24. PMID 33626248
- [Background] van de Leemkolk FEM, Schurink IJ, Dekkers OM, Oniscu GC, Alwayn IPJ, Ploeg RJ, de Jonge J, Huurman VAL. Abdominal Normothermic Regional Perfusion in Donation After Circulatory Death: A Systematic Review and Critical Appraisal. Transplantation. 2020 Sep;104(9):1776-1791. doi: 10.1097/TP.0000000000003345. PMID 32541563